CLINICAL TRIAL: NCT05009693
Title: The Effect of White Light on Fatigue Levels in Patients With Gynecological Cancer: A Double Blind Randomized Trial
Brief Title: Effect of White Light on Fatigue Levels in Patients With Gynecological Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Burcu Tuncer Yilmaz, Phd Research Assistant, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WHITELTESOGU
Record Dates: First submitted 2021-08-02; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Cancer-related Fatigue; Light; Therapy, Complications
Keywords: Cancer-related fatigue; White light therapy; Chemotherapy; Clinical trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- white light intervention group (Experimental): Between the second and the eighth days of the application phase, the patients in the intervention group were administered a standard white light at 10,000 Lux intensity by an independent nurse (RA1) in their home environment using a Litebook Elite light source (The Litebook Company Ltd., Medicine Hat, AB). The distance between the light source and the patient's face was set at 50 cm, and the intensity of the light for each patient was checked using a Lux Meter. The intervention was applied between 07:00 and 10:00 in the morning for 30 minutes without interruption, and it was continued for seven successive days. The light application procedure was followed based on the previous studies on oncology patients. The second and third evaluations of the fatigue status of patients were completed on the 9th and 21st days.
  Interventions: Other: White Light Application
- Control group (No Intervention)

INTERVENTIONS:
Other: White Light Application — White Light Therapy
  Arms: white light intervention group

SUMMARY:
White light therapy is one of the non-pharmacological methods in the management of fatigue. Cancer-related fatigue (CRF) is a persistent, subjective sense of physical, emotional, and/or cognitive tiredness or burnout. It is associated with cancer or cancer treatment from the first diagnosis until the end of life that is not proportional to recent physical activity.

It was founded that 10,000 Lux bright white light administered in the morning hours reduced fatigue by 17% in patients with cancer and that the mean fatigue scores of patients decreased from 30.37 to 9.48 compared to before the light administration. According to NCCN (2020), white light of 10,000 Lux can be applied for 30-90 minutes in the morning hours to regulate sleep and manage fatigue in the post treatment period as well as in cancer patients receiving active treatment. However, studies on this subject consist of small sample groups, and more studies are needed to identify the risks and benefits of the application and to determine the optimal application time and duration. The present study was aimed to evaluate the effect of white light on the fatigue levels of patients with gynecological cancer who were treated with chemotherapy. The patients with high levels of fatigue in every dimension were selected so as to have a homogeneous group. The research hypotheses were determined as follows:

H0: White light has no effect on fatigue levels in patients with gynecological cancer.

H1: White light reduces fatigue levels in patients with gynecological cancer.

ELIGIBILITY:
Inclusion Criteria:

* had a normal state of consciousness,
* had no communication disorders, did not work in the night shift,
* had a general fatigue level score of ≥1 according to the Brief Fatigue Inventory

Exclusion Criteria:

* had natural/artificial lenses,
* used medication that causes photosensitivity (tetracycline, doxycycline, nalidixic acid, voriconazole, amiodarone, hydrochlorothiazide, naproxen, piroxicam, chlorpromazine)
* had a change in their treatment plan in the last 6 weeks were not included in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
White light changes general fatigue scores | general fatigue levels of patients on 0., 9. and 21. days
  White light changes general fatigue levels in patients with gynecological cancer

SECONDARY OUTCOMES:
White light changes activity fatigue scores | activity fatigue levels of patients on 0., 9. and 21. days
  White light changes activity fatigue levels in patients with gynecological cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University Faculty of Medicine, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson JA, Subnis U, Carlson LE, Garland SN, Santos-Iglesias P, Piedalue KL, Deleemans JM, Campbell TS. Effects of a light therapy intervention on diurnal salivary cortisol in fatigued cancer survivors: A secondary analysis of a randomized controlled trial. J Psychosom Res. 2020 Dec;139:110266. doi: 10.1016/j.jpsychores.2020.110266. Epub 2020 Oct 6. PMID 33070045
- [Background] National Comprehensive Cancer Network (NCCN). Clinical Practice Guidelines in Oncology. Cancer related fatigue [Internet]. Version 1.2021. 2020. Available from: https://www.nccn.org/professionals/physician_gls/pdf/fatigue.pdf
- [Background] Fabi A, Bhargava R, Fatigoni S, Guglielmo M, Horneber M, Roila F, Weis J, Jordan K, Ripamonti CI; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Cancer-related fatigue: ESMO Clinical Practice Guidelines for diagnosis and treatment. Ann Oncol. 2020 Jun;31(6):713-723. doi: 10.1016/j.annonc.2020.02.016. Epub 2020 Mar 12. No abstract available. PMID 32173483
- [Background] Nautiyal V, Lal P, Verma M, Yadav R, Singh N, Kumar S. Evaluation of fatigue in head and neck cancer patients undergoing (intensity modulated radiation therapy) radiotherapy: a prospective study. Asian J Oncol. 2015;1(1).
- [Background] Berger AM, Kuhn BR, Farr LA, Von Essen SG, Chamberlain J, Lynch JC, Agrawal S. One-year outcomes of a behavioral therapy intervention trial on sleep quality and cancer-related fatigue. J Clin Oncol. 2009 Dec 10;27(35):6033-40. doi: 10.1200/JCO.2008.20.8306. Epub 2009 Nov 2. PMID 19884558
- [Background] Nowe E, Friedrich M, Leuteritz K, Sender A, Stobel-Richter Y, Schulte T, Hinz A, Geue K. Cancer-Related Fatigue and Associated Factors in Young Adult Cancer Patients. J Adolesc Young Adult Oncol. 2019 Jun;8(3):297-303. doi: 10.1089/jayao.2018.0091. Epub 2019 Feb 20. PMID 30789284
- [Background] Prue G, Allen J, Gracey J, Rankin J, Cramp F. Fatigue in gynecological cancer patients during and after anticancer treatment. J Pain Symptom Manage. 2010 Feb;39(2):197-210. doi: 10.1016/j.jpainsymman.2009.06.011. Epub 2009 Dec 7. PMID 19995675
- [Background] Partridge AH, Jacobsen PB, Andersen BL. Challenges to Standardizing the Care for Adult Cancer Survivors: Highlighting ASCO's Fatigue and Anxiety and Depression Guidelines. Am Soc Clin Oncol Educ Book. 2015:188-94. doi: 10.14694/EdBook_AM.2015.35.188. PMID 25993156
- [Background] Alcantara-Silva TR, de Freitas-Junior R, Freitas NMA, de Paula Junior W, da Silva DJ, Machado GDP, Ribeiro MKA, Carneiro JP, Soares LR. Music Therapy Reduces Radiotherapy-Induced Fatigue in Patients With Breast or Gynecological Cancer: A Randomized Trial. Integr Cancer Ther. 2018 Sep;17(3):628-635. doi: 10.1177/1534735418757349. Epub 2018 Apr 10. PMID 29633652
- [Background] Howell D, Keller-Olaman S, Oliver TK, Hack TF, Broadfield L, Biggs K, Chung J, Gravelle D, Green E, Hamel M, Harth T, Johnston P, McLeod D, Swinton N, Syme A, Olson K. A pan-Canadian practice guideline and algorithm: screening, assessment, and supportive care of adults with cancer-related fatigue. Curr Oncol. 2013 Jun;20(3):e233-46. doi: 10.3747/co.20.1302. PMID 23737693
- [Background] Starreveld DEJ, Daniels LA, Valdimarsdottir HB, Redd WH, de Geus JL, Ancoli-Israel S, Lutgendorf S, Korse CM, Kieffer JM, van Leeuwen FE, Bleiker EMA. Light therapy as a treatment of cancer-related fatigue in (non-)Hodgkin lymphoma survivors (SPARKLE trial): study protocol of a multicenter randomized controlled trial. BMC Cancer. 2018 Sep 10;18(1):880. doi: 10.1186/s12885-018-4746-2. PMID 30200906
- [Background] Johnson JA, Garland SN, Carlson LE, Savard J, Simpson JSA, Ancoli-Israel S, Campbell TS. Bright light therapy improves cancer-related fatigue in cancer survivors: a randomized controlled trial. J Cancer Surviv. 2018 Apr;12(2):206-215. doi: 10.1007/s11764-017-0659-3. Epub 2017 Nov 10. PMID 29127575
- [Background] Mendoza TR, Wang XS, Cleeland CS, Morrissey M, Johnson BA, Wendt JK, Huber SL. The rapid assessment of fatigue severity in cancer patients: use of the Brief Fatigue Inventory. Cancer. 1999 Mar 1;85(5):1186-96. doi: 10.1002/(sici)1097-0142(19990301)85:53.0.co;2-n. PMID 10091805
- [Background] Redd WH, Valdimarsdottir H, Wu LM, Winkel G, Byrne EE, Beltre MA, Liebman ES, Erazo T, Hayes JA, Isola L, Scigliano E, Meschian Y, Lutgendorf S, Ancoli-Israel S. Systematic light exposure in the treatment of cancer-related fatigue: a preliminary study. Psychooncology. 2014 Dec;23(12):1431-4. doi: 10.1002/pon.3553. Epub 2014 May 2. No abstract available. PMID 24798589
- [Background] Steur LMH, Kaspers GJL, Van Someren EJW, Van Eijkelenburg NKA, Van der Sluis IM, Dors N, Van den Bos C, Tissing WJE, Grootenhuis MA, Van Litsenburg RRL. Sleep-wake rhythm disruption is associated with cancer-related fatigue in pediatric acute lymphoblastic leukemia. Sleep. 2020 Jun 15;43(6):zsz320. doi: 10.1093/sleep/zsz320. PMID 31889198
- [Background] Kronish IM, Cheung YK, Julian J, Parsons F, Lee J, Yoon S, Valdimarsdottir H, Green P, Suls J, Hershman DL, Davidson KW. Clinical Usefulness of Bright White Light Therapy for Depressive Symptoms in Cancer Survivors: Results from a Series of Personalized (N-of-1) Trials. Healthcare (Basel). 2019 Dec 30;8(1):10. doi: 10.3390/healthcare8010010. PMID 31905890
- [Derived] Ozerdogan N, Ozkaraman A, Tuncer Yilmaz B, Oge T, Yalcin OT. The Effect of Bright White Light on Fatigue Levels in Patients with Gynecological Cancer: A Randomized Control Trial. J Palliat Care. 2023 Oct;38(4):416-423. doi: 10.1177/08258597221127795. Epub 2022 Sep 25. PMID 36154518

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT05009693/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT05009693/ICF_001.pdf